CLINICAL TRIAL: NCT05613192
Title: The Effect of High Oral Loading Dose of Cholecalciferol in Non-Alcoholic Fatty Liver Disease Patients. A Randomized Placebo Controlled Trial
Brief Title: Effectiveness of Inactive Vitamin D Supplementation in Non-Alcoholic Fatty Liver Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Maher Abd El Kader El Borolossy, Lecturer of clinical pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NHTMRI-IRB 10-22
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: non-alcoholic fatty liver- vitamin D
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Group 1: patients received the standard conventional therapy in addition to placebo for 4 months.
  Group 2: patients received the standard conventional therapy in addition to a single oral dose of cholecalciferol 300,000 IU followed by oral cholecalciferol 800 IU daily for 4 months.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study medications were given to the patients by an unblinded pharmacist to ensure the right treatment assignment, however this pharmacist was not included in the outcome assessment.
  All patients were diagnosed with NAFLD depending on abdominal ultrasonography performed by a radiologist where the liver brightness and liver parenchyma with diffuse echogenicity in confirm the diagnosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): Group 1: patients receive the standard conventional therapy in addition to placebo for 4 months.
  Interventions: Drug: Cholecalciferol
- Cholecalciferol (Experimental): Group 2: patients receive the standard conventional therapy in addition to a single oral dose of cholecalciferol 300,000 IU followed by oral cholecalciferol 800 IU daily for 4 months.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — patients receive the standard conventional therapy in addition to a single oral dose of cholecalciferol 300,000 IU followed by oral cholecalciferol 800 IU daily for 4 months.
  Other Names: native vitamin D

SUMMARY:
Aim of work The aim of our study is to assess the effectiveness and safety of high oral loading dose of inactive vitamin D supplementation on the clinical parameters related to liver steatosis, glycaemic control, insulin resistance and metabolic profile in NAFLD patients

DETAILED DESCRIPTION:
Aim of work The aim of our study is to assess the effectiveness and safety of high oral loading dose of inactive vitamin D supplementation on the clinical parameters related to liver steatosis, glycaemic control, insulin resistance and metabolic profile in NAFLD patients

Patients and Methods The present study is prospective, simply (via computer generated sequence) randomized controlled double blinded study, will be conducted on NAFLD patients in the outpatient liver clinics of EL Sahel Teaching hospital, Cairo, Egypt, Inclusion criteria: To be included in the study, patients have to fulfil the following inclusion criteria: male or female patients >19 years of age; presence of fatty liver detected by upper abdominal ultrasound echography (US) and with diagnosis of T2D according to ADA 2019 criteria.

Exclusion Criteria: The main exclusion criteria from the study are as follows: Pregnancy and lactation, history of alcohol abuse (as defined by an average daily consumption of alcohol > 30 g/day in men and > 20 g/day women), cirrhosis, autoimmune hepatitis and other causes of liver disease (viral hepatitis, hemochromatosis, Wilson's disease), drug induced hepatitis, chronic enteropathies, Chronic kidney disease, hyper/hypoparathyroidism, known hypersensitivity to cholecalciferol.

Hundred eligible patients will be included into the study and randomized by simple randomization into either of the 2 groups:

Group 1: 50 patients receive the standard conventional therapy in addition to placebo for 4 months.

Group 2: 50 patients receive the standard conventional therapy in addition to a single oral dose of cholecalciferol 300,000 IU followed by oral cholecalciferol 800 IU daily for 4 months.

The following laboratory tests will be measured: a- Glycaemic control: Fasting blood glucose (FBG mg/dl), glycated haemoglobin (HbA1C%), Fasting insulin (mU/L), Insulin resistance index calculated by the homeostasis model assessment insulin resistance (HOMA-IR) method using the product of fasting insulin and fasting plasma glucose divided by 405. The cut off value of HOMA-IR is more than 1.64.

b-Liver function tests: Alanine transaminase (ALT U/L), Aspartate transaminase (AST U/L), Albumin (g/dl), Gamma glutamyl transferase (GGT U/L), Alkaline phosphatase (ALP U/L).

c- Lipid Profile: Low density lipoprotein (LDL-C mg/dl), High density lipoprotein (HDL-C mg/dl), Triglycerides (TG mg/dl), Total cholesterol (TC mg/dl) d- Other markers: High sensitivity C reactive protein (hsCRP mg/dl), Alfa fetoprotein (AFP ng/ml), serum 25-hydroxy vitamin D (25(OH) D ng/ml) All Patients were followed up every 2 weeks by the clinical pharmacist in charge through patient encounter to ensure the compliance to the treatment regimen and to assess any adverse side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years with fatty liver diagnosis by using upper abdominal ultrasound echography (US)
* patients with T2D diagnosed according to ADA 2019 criteria and treated with metformin.

Exclusion Criteria:

* Pregnant and/or lactating women,
* excessive alcohol use (as defined by an average daily consumption of alcohol > 30 g/day in men and > 20 g/day women),
* patients with other causes of chronic liver disease as viral hepatitis, drug induced hepatitis, autoimmune hepatitis, patients suffering of chronic kidney disease, hyper/hypoparathyroidism,
* hypersensitivity to cholecalciferol,
* hypercalcemia,
* patients taking supplementation with vitamin D,
* calcium and medications affecting calcium/vitamin D metabolism (as: anticonvulsants, glucocorticoids, antacids).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of cholecalciferol on glycaemic control parameters in non alcoholic fatty liver disease | at Baseline and at week 16
  Decrease in glycated haemoglobin in NAFLD patients

SECONDARY OUTCOMES:
Efficacy of cholecalciferol on the degree of steatosis in non alcoholic fatty liver disease | at Baseline and at week 16
  Decrease in the degree of steatosis imaged by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Radwa El Borolossy, Principal Investigator — Faculty of pharmacy Ain Shams university
Locations (1):
- National hepatology and tropical medicine research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed AA, Halim AA, Mohamed S, Mahmoud SM, Bahgat Eldemiry EM, Mohamed RS, Shaheen MM, Naguib GG, Muharram NM, Khalil MG, Saed S, Ibrahim R, Salah Seif A, Kamal N, Nasraldin K, Abdelrahman AE, El Borolossy R. The effect of high oral loading dose of cholecalciferol in non-alcoholic fatty liver disease patients. A randomized placebo controlled trial. Front Pharmacol. 2023 Mar 14;14:1149967. doi: 10.3389/fphar.2023.1149967. eCollection 2023. PMID 36998617